CLINICAL TRIAL: NCT06646224
Title: A Clinical Trial to Evaluate the Efficacy and Safety of the CorVad Percutaneous Ventricular Assist System in the Treatment of Cardiogenic Shock Caused by Cardiomyopathy
Brief Title: Efficacy and Safety of the CorVad Percutaneous Ventricular Assist System in Cardiogenic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_Corvad_CMCS
Record Dates: First submitted 2024-10-08; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CorVad Percutaneous Ventricular Assist System (Experimental): Subjects with cardiogenic shock caused by cardiomyopathy will be supported by the CorVad Percutaneous Ventricular Assist System
  Interventions: Device: CorVad Percutaneous Ventricular Assist System

INTERVENTIONS:
Device: CorVad Percutaneous Ventricular Assist System — The CorVad Percutaneous Ventricular Assist System provides circulatory support for patients with cardiogenic shock.

SUMMARY:
This study aims to evaluate the safety and effectiveness of the CorVad Percutaneous Ventricular Assist System for providing circulatory support in patients with cardiogenic shock caused by cardiomyopathy. This will be assessed through a prospective, multicenter, single-arm clinical trial involving patients with cardiogenic shock. The focus will be on determining the device's ability to improve survival outcomes and reduce the risk of related adverse events in these patients.

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm clinical trial of the CorVad Percutaneous Ventricular Assist System is designed to measure the survival rate of subjects. The survival rate is defined as follows:

* 1. Recovery: Survival at 30 days post-device removal or at discharge (whichever is longer);
* 2. Bridge to Other Therapy: Survival at 30 days post-heart transplantation or left ventricular assist device (LVAD) implantation.

The study plans to enroll 50 subjects. The target population consists of patients with cardiogenic shock caused by cardiomyopathy who provide informed consent through a form approved by the Ethics Committee (EC). Subjects who meet the enrollment criteria, as determined by the investigator, will receive the trial device in accordance with study requirements and will be followed up to assess the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of subjects must be between 18 and 80 years old (inclusive).
* 2. Presence of heart failure or cardiac dysfunction caused by cardiomyopathy.
* 3. Occurrence of cardiogenic shock under adequate blood volume, which must meet one of the following conditions:

  1. Rapidly Worsening Cardiogenic Shock: Progressive hemodynamic instability requiring repeated administration of vasopressors to maintain mean arterial pressure >50 mmHg, and left ventricular systolic function is impaired (LVEF <35% or LVEF 35-55% with significant mitral regurgitation).
  2. Severe Cardiogenic Shock: Cardiac index (CI) < 2.2 L/min/m² + norepinephrine dose > 0.1 µg/kg/min + dopamine or dobutamine dose > 10 µg/kg/min; systolic blood pressure < 90 mmHg + norepinephrine dose > 0.2 µg/kg/min + dopamine or dobutamine dose > 10 µg/kg/min + LVEF < 35% or LVEF 35-55% with significant mitral regurgitation.
* 4. Two consecutive blood lactate measurements ≥ 3.0 mmol/L (with at least a 30-minute interval).
* 5. The subject or their guardian must be able to understand the purpose of the trial, sign the informed consent form, demonstrate good compliance after discharge, and be willing to complete clinical follow-up.

Exclusion Criteria:

* 1. Continuous cardiopulmonary resuscitation (CPR) cannot restore circulation.
* 2. CorVad cannot be implanted or applied (including but not limited to left ventricular mural thrombus, presence of artificial aortic valve or cardiac contraction devices, moderate to severe aortic stenosis, moderate to severe aortic regurgitation, aortic dissection, aneurysm, or severe abnormalities of the ascending aorta and/or aortic arch, blood cell fragility, or hemolytic blood disorders).
* 3. Inability to use heparin for anticoagulation therapy.
* 4. Shock caused by other reasons (e.g., myocardial infarction, arrhythmia, hypovolemia, septic shock, etc.).
* 5. Presence of unrepaired cardiac structural damage (e.g., chordal rupture, ventricular septal perforation, free wall rupture, etc.).
* 6. Severe right heart failure.
* 7. Pregnant or breastfeeding women.
* 8. Currently participating in another clinical trial of a drug or device that has not yet reached its primary endpoint.
* 9. Any other circumstances deemed inappropriate for inclusion in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-12 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of Subjects | Recovery: 30 days post-CorVad removal or discharge (which is longer); Bridge to Other Therapy: 30 days post-heart transplantation or LVAD implantation
  Survival is defined as:
  1. Recovery: Survival at 30 days post device removal or at discharge (whichever is longer);
  2. Bridge to Other Therapy: Survival at 30 days post heart transplantation or left ventricular assist device (LVAD) implantation.

SECONDARY OUTCOMES:
In-Hospital Mortality Rate | 30 days post-CorVad removal or discharge (which is longer)
14-Day Mortality Rate After CorVad Removal | 14 days post-CorVad removal
Stroke | Within 30 days post-CorVad removal
Cardiovascular-Cause Mortality | Within 30 days post-CorVad removal
Re-Hospitalization Due to Cardiovascular Reasons | Within 30 days post-CorVad removal
  Re-hospitalization for cardiovascular disease
MCS-ARC Type 3, 4, 5 Bleeding | Within 30 days post-CorVad removal
Serious Device-Related Adverse Events | Within 30 days post-CorVad removal
  Serious device-related adverse events include but are not limited to cardiac structural damage, severe limb ischemia (pallor, pulselessness, and necrosis), puncture site infection, acute kidney injury, arrhythmias requiring cardiopulmonary resuscitation, damage to the aorta and aortic valve, hemolysis resulting in subject death, permanent or serious disability, significantly prolonged hospital stay, or surgical intervention required.
Duration of Device Use | Recovery: 30 days post-CorVad removal or discharge (which is longer); Bridge to Other Therapy: 30 days post-heart transplantation or LVAD implantation
Device Malfunction | During CorVad operation
  Device malfunction is defined as a flow rate of less than 1L/min at S5 or higher speed level lasting more than 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences.Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
At this moment the IPD is not yet available for access and will be updated when it is ready.